CLINICAL TRIAL: NCT03069092
Title: Comparison of the Cardiovascular Benefits of Resistance, Aerobic, and Combined Exercise
Acronym: CardioRACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iowa State University (Other)
Responsible Party: Principal Investigator, Duck-chul Lee, Assistant Professor, Iowa State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01HL133069-01 (NIH)
Record Dates: First submitted 2017-02-23; First posted 2017-03-03 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Exercise; Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Aerobic exercise (AE) (Experimental): AE training will consist of 60 min of treadmill, elliptical, or bike exercise at a moderate to vigorous intensity (50-80% of heart rate reserve). Intensity of the exercise sessions will be built up gradually. Sessions will occur 3 times per week for the duration of the 1 year trial.
  Interventions: Behavioral: aerobic exercise
- Resistance exercise (RE) (Experimental): RE will consist of 3 sets of 8-15 repetitions at 50-80% of 1 rep-max of each exercise for 12 exercises (chest press, shoulder press, pull-down, back extension, abdominal crunch, torso rotation, biceps curl, triceps extension, leg press, leg extension, leg curl, and calf raise). Weight loads will be increased gradually. With one minute of rest between sets, this plan is estimated to take approximately 60 minutes per session. Sessions will occur 3 times per week for the duration of the 1 year trial.
  Interventions: Behavioral: resistance exercise
- Combined Resistance and Aerobic Exercise (Experimental): Participants will perform exactly the same AE and RE exercises as listed previously; however, the time of AE and RE will each be reduced to 30 min (for 60 min/session total). For the RE aspect, participants will perform 2 sets of 8-15 repetitions of 9 exercises (excluding biceps curl, triceps extension, and calf raise, as these are minor muscle groups). Exercise intensity and resistance will be increased gradually. Combined AE and RE sessions will take place 3 times per week for the duration of the trial.
  Interventions: Behavioral: Combined resistance and aerobic exercise
- No training control (No Intervention): Participants in this group will be asked to maintain their current level of activity during the 1 year study period. After 1 year, they will be offered the training program of their choice (AE, RE, or combined).

INTERVENTIONS:
Behavioral: aerobic exercise — AE training will consist of 60 min of treadmill, elliptical, or bike exercise at a moderate to vigorous intensity (50-80% of heart rate reserve). Intensity of the exercise sessions will be built up gradually. Sessions will occur 3 times per week for the duration of the 1 year trial.
  Arms: Aerobic exercise (AE)
Behavioral: resistance exercise — RE will consist of 3 sets of 8-15 repetitions at 50-80% of 1 rep-max of each exercise for 12 exercises (chest press, shoulder press, pull-down, back extension, abdominal crunch, torso rotation, biceps curl, triceps extension, leg press, leg extension, leg curl, and calf raise). Weight loads will be increased gradually. With one minute of rest between sets, this plan is estimated to take approximately 60 minutes per session. Sessions will occur 3 times per week for the duration of the 1 year trial
  Arms: Resistance exercise (RE)
Behavioral: Combined resistance and aerobic exercise — Participants will perform exactly the same AE and RE exercises as listed previously; however, the time of AE and RE will each be reduced to 30 min (for 60 min/session total). For the RE aspect, participants will perform 2 sets of 8-15 repetitions of 9 exercises (excluding biceps curl, triceps extension, and calf raise, as these are minor muscle groups). Exercise intensity and resistance will be increased gradually. Combined AE and RE sessions will take place 3 times per week for the duration of the trial.
  Arms: Combined Resistance and Aerobic Exercise

SUMMARY:
As the leading cause of death, cardiovascular disease (CVD) accounts for about one-third of U.S. mortality. Physical inactivity, one of the main CVD risk factors, causes 6% of coronary heart disease worldwide. The American Heart Association has identified cardiovascular health behaviors including smoking, obesity, diet, and aerobic exercise; however, resistance exercise was not included due to the limited evidence of its efficacy. Comparatively, the cardiovascular benefits of aerobic training have been well-documented whereas the independent and additive benefits of resistance training on cardiovascular health have not been established. Thus, this project is aimed to answer one of the most common questions about exercise and health:"What type or combination of exercise is most effective for CVD prevention?" This project will significantly contribute to developing more effective CVD prevention approaches, advancing more comprehensive physical activity guidelines, and providing important insights and novel opportunities for the future science of physical activity and health.

DETAILED DESCRIPTION:
Participants will be randomly assigned to aerobic exercise, resistance exercise, combined aerobic and resistance exercise, or a no exercise control group for 1 year. Participants in all four groups will receive healthy diet and lifestyle education sessions and will track their daily steps, body weights, and food intake throughout the 1-year intervention. They will also complete baseline, 6-month, and 12-month physical examinations, which will include assessments of blood pressure, blood lipids, body composition, and aerobic and muscular fitness.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker
* Systolic/diastolic blood pressure of 120-139/80-89 mmHg (without taking any anti-hypertensive medication)
* Overweight or obese: body mass index of 25-40 kg/m2; Asian 23-40 kg/m2
* Inactive: less than 150 min/week of exercise over the past 3 months
* Capable of performing the required exercise training

Exclusion Criteria:

* Unstable coronary heart disease or heart failure
* Uncontrolled arrhythmias or severe aortic stenosis
* Acute myocarditis, endocarditis, or pericarditis
* Cancer, requiring treatment in the past 5 years
* Autoimmune diseases, affecting the immune system
* Plans to be away/travel for greater than 4 weeks in the next year
* Pregnancy/anticipated pregnancy during the study
* Other medical condition that is life-threatening or can interfere with or be aggravated by the exercise training

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Change in composite cardiovascular disease risk score (z-score) | 12 months
  The primary outcome is the change from baseline in the composite cardiovascular disease risk score (z-score) calculated using resting blood pressure, low-density lipoprotein cholesterol, fasting glucose, and percent body fat. Each risk factor will be individually standardized and expressed as sex-specific z-score by using the formula = (value - mean)/standard deviation for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Duck-chul Lee, Ph.D., Principal Investigator — Iowa State University
Locations (1):
- Iowa State University, Ames, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Datasets will be available to outside researchers and public health professionals through the web sites of the ClinicalTrials.gov and The Physical Activity Epidemiology Laboratory at Iowa State University. Outside researchers can learn what data are available and request a de-identified dataset (stripped of all personal health identifiers). All outside investigators must pass an NIH-approved equivalent course on the Protection of Human Subjects. All data requests will be discussed with the research team and approval will be obtained from the institutional review board overseeing the proposal of the data analysis project. Findings from the proposed study will also be disseminated at national and international meetings and publish the findings in peer-reviewed journals. The investigators seek to maximize the knowledge discovered from this study by sharing data to expedite the translation of research into practice to improve cardiovascular health.

REFERENCES:
- [Derived] Brellenthin AG, Lanningham-Foster LM, Kohut ML, Li Y, Church TS, Blair SN, Lee DC. Comparison of the Cardiovascular Benefits of Resistance, Aerobic, and Combined Exercise (CardioRACE): Rationale, design, and methods. Am Heart J. 2019 Nov;217:101-111. doi: 10.1016/j.ahj.2019.08.008. Epub 2019 Aug 15. PMID 31520895
- See also: Information regarding Dr. Lee's laboratory at Iowa State University. — http://www.kin.hs.iastate.edu/research/physical-activity-epidemiology/
- See also: Study website, including contact information for recruitment — https://research.hs.iastate.edu/cardiorace

DOCUMENTS (1):
  • Informed Consent Form (2019-03-05): https://cdn.clinicaltrials.gov/large-docs/92/NCT03069092/ICF_000.pdf